CLINICAL TRIAL: NCT05136781
Title: Assessment of DEXAMETHASONE to Prevent Respiratory Complications After Non Urgent Thoracic Surgery
Brief Title: DEXAMETHASONE for Non-urgent Thoracic Surgery
Acronym: SURTHODEX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0202
Record Dates: First submitted 2021-11-16; First posted 2021-11-29 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Thoracic Surgery; Anesthesiology; Corticosteroids; Respiratory Complication
Keywords: Thoracic surgery; Anesthesiology; Corticosteroids; Respiratory Complication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thoracic surgery is at high risk of respiratory complications. Despite the improvement of surgical procedures such as video-thoracoscopy, respiratory complications appear in 15 to -20% of procedures. Thoracic surgery induces local pulmonary inflammation which is involved in the occurrence of post-operative respiratory failure. Similarly to the example of the acute respiratory distress syndrome, corticosteroids could reduce lung injury secondary to immunological stress. In addition, recent studies suggest that dexamethasone could lead to a reduction of respiratory complications after major non cardiothoracic surgery.

Since dexamethasone is recommended to prevent postoperative nausea and vomiting, around one in two patients receive dexamethasone during anesthetic induction. By retrospective analysis with compensation of bias by propensity score, the investigators aim to assess the effect of dexamethasone to prevent respiratory complications

ELIGIBILITY:
Inclusion Criteria:

* age : minimum 18 years old
* Patients who underwent scheduled lung resection surgery

Exclusion Criteria:

* absence of patient's consent
* age under 18 years
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent scheduled lung resection surgery
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
incidence of respiratory failure rates between patients receiving or not DEXAMETHASONE | 7 days following surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No